CLINICAL TRIAL: NCT02434237
Title: Robot-Aided Neurorehabilitation of the Upper Extremities
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK 04 2005
Record Dates: First submitted 2014-10-13; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Robot-aided Arm Therapy, Brain Injury, Motor Relearning Programme, Activities of Daily Living
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients
- healthy subjects

SUMMARY:
Task-oriented repetitive movement can improve movement performance in patients with neurological or orthopedic lesions. The application of robotics can serve to assist, enhance, evaluate, and document neurological and orthopedic rehabilitation of movements. Arm therapy is used in neurological rehabilitation for patients with paralyzed upper extremities due to lesions of the central or peripheral nervous system, e.g. after stroke or spinal cord injury. The goal of the therapy is to recover motor function, improve movement coordination, learn new motion strategies ("trick movements"), and/or prevent secondary complications such as muscle atrophy, osteoporosis, and spasticity.

ELIGIBILITY:
Inclusion Criteria:

Patients with neurological disability of the upper limb with qualification for arm training, e.g. after stroke and spinal cord injury

Exclusion Criteria:

* limitations of the join mobility
* osteoporosis
* cardiovascular disease
* injury of the upper limb
* decubitus
* psychic diseases (like schizophrenia, dementia, depression)
* Body weight > 120kg
* pacemaker.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and neurological patients after stoke or spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2005-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The acceptanece of the arm rehabilitation robot therapy and the influence to the motivation through the visual feedback. | A measure lasts approx. 90 minutes. Every participant once.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Swiss Federal Institute of Technology, Zurich, Canton of Zurich, Switzerland